CLINICAL TRIAL: NCT02645734
Title: The Comparison Between the Therapeutic Effect of Intravitreal Bevacizumab and Ziv-aflibercept in Diabetic Macular Edema
Brief Title: The Effect of Bevacizumab and Ziv-aflibercept in Diabetic Macular Edema
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Assistant Professor of Ophthalmology, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 93210
Record Dates: First submitted 2016-01-02; First posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-10

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Bevacizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Injection intravitreous bevacizumab (Active Comparator): Injection intravitreous bevacizumab at a dose 1.25mg
  Interventions: Drug: bevacizumab
- Injection ziv-aflibercept at dose of 1.25 mg (Active Comparator): Injection ziv-aflibercept at dose of 1.25 mg
  Interventions: Drug: ziv-aflibercept 1.25 mg
- Injection ziv-aflibercept at dose of 2.5 mg (Active Comparator): Injection ziv-aflibercept at dose of 2.5 mg
  Interventions: Drug: ziv-aflibercept 2.5mg

INTERVENTIONS:
Drug: bevacizumab — 1.25 mg of bevacizumab is injected
  Arms: Injection intravitreous bevacizumab
Drug: ziv-aflibercept 1.25 mg — 1.25 mg of ziv-aflibercept is injected
  Arms: Injection ziv-aflibercept at dose of 1.25 mg
Drug: ziv-aflibercept 2.5mg — 2.5 mg of ziv-aflibercept is injected
  Arms: Injection ziv-aflibercept at dose of 2.5 mg

SUMMARY:
In this double clinical trial 132 patient with the history of DME (Diabetic Macular Edema) to receive intravitreous bevacizumab at a dose of 1.25mg (44 patient) , ziv-aflibercept at dose of 1.25 mg (44 patient) , ziv-aflibercept at dose of 2.5 mg (44 patient) .

The study drugs were administered as often as every 4 weeks for 3 months.monitoring of best-corrected visual acuity, CST ( Central Subfield Thickness) by OCT (Optical coherence tomography) was done from base line ,4 weeks, 8weeks after injection.

ELIGIBILITY:
Inclusion Criteria:

* The patient at least 18 years old had type 1 or 2 diabetes who presented with Central DME involvement (defined as retinal thickening involving 1mm central sub field thickness(CCT)
* Have at least a BCVA ( best corrected visual acuity) between 20/50 to 20/320 Snellen equivalent
* Have received to anti-VEGF( anti -vascular endothelial growth factor) and laser treatment within the previous 3 months

Exclusion Criteria:

* Uncontrolled glaucoma/uncontrolled diabet , high risk PRP(pan-retinal photocoagulation), one eye
* Prior treatment with intravitreal or peribulbar injection and laser therapy during the last 3 months
* Substantial cataract, history of uveitis
* Macular edema due to a cause other than DME
* VMT(Vitreomacular traction ) and ERM (epiretinal membrane)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Primary Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
visual acuity | until 6 month

SECONDARY OUTCOMES:
central subfield thickness(CCT) | until 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Islamic Republic of Iran, Tehran, Iran